CLINICAL TRIAL: NCT01757379
Title: Evaluation of the Bioavailability and Production of Short Chain Fatty Acids in the Colon. A Stable Isotope Study in Healthy Humans.
Brief Title: Determination of the Bioavailability of Short Chain Fatty Acids in Healthy Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor K. Verbeke, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: ML5768
Record Dates: First submitted 2012-12-21; First posted 2012-12-28 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Short Chain Fatty Acids Bioavailability
Keywords: Short chain fatty acids; Acetate; Propionate; Butyrate; Bioavailability
MeSH Terms: interventions — Inulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 13C-labeled acetate (Experimental)
  Interventions: Dietary Supplement: 13C-labeled Acetate
- 13C-labeled propionate (Experimental)
  Interventions: Dietary Supplement: 13C-labeled propionate
- 13C-labeled butyrate (Experimental)
  Interventions: Dietary Supplement: 13C-labeled butyrate
- Inulin (Experimental)
  Interventions: Dietary Supplement: Inulin

INTERVENTIONS:
Dietary Supplement: 13C-labeled Acetate — 400 mg of sodium acetate 1-13C (2 colon delivery capsules with 200 mg)
  Arms: 13C-labeled acetate
Dietary Supplement: 13C-labeled propionate — 340 mg of sodium propionate 1-13C (2 colon delivery capsules with 170 mg)
  Arms: 13C-labeled propionate
Dietary Supplement: 13C-labeled butyrate — 990 mg sodium butyrate 1-13C (2 colon delivery capsules with 495 mg)
  Arms: 13C-labeled butyrate
Dietary Supplement: Inulin — 15 g of inulin dissolved in 200 ml of water
  Arms: Inulin

SUMMARY:
The purpose of the study is to evaluate the bioavailability of acetate, propionate and butyrate in healthy humans using a stable isotope technology.

In addition the level of acetate, propionate and butyrate production from inulin will be determined using the principle of isotope dilution.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Regular dietary pattern (3 meals/day)
* Age: 18-65y
* BMI: 18,5-27 kg/m2

Exclusion Criteria:

* Intake of antibiotics 1 month prior to the study
* Abdominal surgery in the past, with the exception of appendectomy
* Intake of medication influencing the gastro-intestinal system 14 days prior to the study
* In treatment at a dietician
* Intake of pre- and/or probiotics
* Exposure to radioactivity 1 year prior to the study
* Serious chronic disease of the gastrointestinal tract
* Use of medication that affects the gastro-intestinal tract during the last 2 weeks prior to the study
* Pregnancy, pregnancy desire or lactation
* Blood donation during the last 3 months prior to the study
* Diabetes (type 1 or 2)
* Aberrant hemoglobin level (Hb) in blood. Normal between 14.0 and 18.0 g/dL for men and between 12.0 and 16.0 g/dL for women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2011-04; Primary Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Concentrations of the short chain fatty acids (acetate, propionate and butyrate) in plasma and urine samples | 12 hours each test day and 4 test days/volunteer
  Participants performed each 4 test days and they were followed each test day for 12 hours, with sample collections at regular time points. Blood samples were collected every hour during the first 4 hours and afterwards every 20 minutes during 8 hours. Urine samples were collected during 24h in different fractions: 0-4h, 4-8h, 8-12h, 12-24h.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Verbeke, Professor, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven/ UZ Leuven, Leuven, Vlaams-Brabant, Belgium